CLINICAL TRIAL: NCT04707378
Title: Navigated Repetitive Transcranial Magnetic Stimulation for Parkinson's Disease With Depression or Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDREC2020181H(R1)
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease; Depression; Cognitive Impairment
Keywords: Parkinson's Disease; rTMS; Depression; Cognitive Impairment; Navigation; Dorsal Prefrontal Cortex
MeSH Terms: conditions — Parkinson Disease; Depression; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active left DLPFC navigated-rTMS (Active Comparator): Each patient will be given 10 treatment sessions per week for 2 weeks (a total of 10 sessions). In each rTMS session, 1200 pulses of stimuli at an intensity of 100% rest motor threshold (RMT) will give over the left DLPFC. Each session is 20 minutes long and will be consisted of 10Hz stimulation trains (active) over the left DLPFC.
  Interventions: Device: repetitive transcranial magnetic stimulation(rTMS)
- sham left DLPFC navigated-rTMS (Sham Comparator): Each patient will be given 10 treatment sessions per week for 2 weeks (a total of 10 sessions). In each rTMS session, 1200 pulses of sham stimuli at an intensity of 100% rest motor threshold (RMT) will give over the left DLPFC. Each session is 20 minutes long and will be consisted of 10Hz stimulation trains (sham) over the left DLPFC.
  Interventions: Device: repetitive transcranial magnetic stimulation(rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation(rTMS) — Each patient will be given 10 treatment sessions per week for 2 weeks (a total of 10 sessions). In each rTMS session, 1200 pulses of stimuli at an intensity of 100% rest motor threshold (RMT) will give over the left DLPFC. Each session is 20 minutes long and will be consisted of 10Hz stimulation trains (active) over the left DLPFC. For sham control rTMS blocks, the coil will be oriented 90◦ away from the scalp so that no pulses perturbed underlying neural tissue.

SUMMARY:
Depressive symptoms are common non-motor symptoms in patients with Parkinson's disease and seriously affect the quality of life and prognosis of patients. Currently, treatment measures for patients with Parkinson's disease with depression are mainly limited to pharmacotherapy, but the side effects of antidepressants and their interaction with anti-Parkinsonian drugs limit the use of pharmacotherapy. Repetitive transcranial magnetic stimulation (rTMS) is a new painless and non-invasive neuromodulation technique that is commonly used in the treatment of depression. As the number of people with Parkinson's disease increases in China, the number of patients with Parkinson's disease and depression requiring rTMS treatment will also increase. The size and shape of individual brains, the distance between the stimulation coil and the responding neuronal tissue, and the location and orientation of anatomical structures are all different, and the use of common localization methods is usually limited by these individual anatomical differences. The traditional method relies on manual positioning of the coil, which is time-consuming and inefficient, and it is difficult to meet the requirements of position, angle, and coil orientation simultaneously. Studies have shown that the benefits of using navigation for rTMS treatment are up to twice as high as those of non-navigation methods. Therefore precise localization is a must for the future standardized application of rTMS in the development of patients with Parkinson's disease with depression. In this study, we applied repetitive transcranial magnetic stimulation with neuronavigation to treat patients with Parkinson's disease and depression, and reconstructed cephalometric models with individual cranial imaging data to individualize and precisely target stimulation sites, making rTMS more precise and effective in treating patients with Parkinson's disease and depression, and providing new avenues for further clinical and scientific research.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients between 18 and 85 years of age with idiopathic PD (diagnosed as "confirmed PD" or "likely PD" according to the 2015 MDS Parkinson's diagnostic criteria), regardless of gender.

  2. Meet the DSM-IV diagnostic criteria for depressive episodes. 3. If there is a combination of anti-Parkinsonian medications, the anti-Parkinsonian medication regimen and dose must remain stable for ≥ 28 days and be maintained at that dose for the duration of treatment.

  4. Not taking any antidepressant medication for the last 2 months. 5. the subject/their legal representative is able to comply with the study protocol and visit schedule.

  6. The patient or his/her legal guardian agrees to participate in this trial and signs an informed consent form.

Exclusion Criteria:

* 1. Secondary Parkinson's syndrome caused by vascular factors, toxins, drugs, etc., or Parkinson's superimposed syndrome.

  2. PD patients with persistent head tremor. 3. Dementia. 4. Patients with suicidal tendencies and psychotic symptoms. 5. Patients with consciousness disorders, history of stroke, severe neurological/psychiatric disorders such as transient ischemic attack and other severe organic diseases within 1 year prior to screening (Visit 1) 6. Have contraindications to rTMS(e.g., implantation of cochlear implants, deep brain stimulation, pacemakers, medical pumps, and other metal-containing devices near stimulation coils; history of epilepsy; history of traumatic brain injury, brain tumor, encephalitis, cerebrovascular disease, cerebral metabolic disease; sleep deprivation, unrecovered jet lag, intoxication, overexertion; pregnancy; severe or recent heart disease, etc.) 7. Have contraindications to MRI scanning (including metal implants, retractors, braces, or claustrophobia).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale（HAMD） | 1 months
  The Hamilton Depression Rating Scale (HAMD) is a 24-item interviewer administered structure questionaire designed to assess symptoms of depression. Items are scored with a range of 0-4, though 11 of the items are scored between 0 and 2. A total score is then calculated of all items which can range from 0 to 74. A higher score is indicative of more depressive symptoms, and a lower score post-tx is indicative of better outcome.
Beck Depression Inventory（BDI） | 1 months
  The Beck Depression Inventory (BDI) is a 21-item self-report questionaire that measures depressive symptoms. Each item is scored on a scale of 0-3, and items are summated to yield a total score. A higher score is indicative of greater symptoms of depression. Total scores may range between 0 and 63. A score greater than or equal of 14 is suggestive of clinically significant symptoms.

SECONDARY OUTCOMES:
Hamilton Anxiety Scale（HAMA） | 1 months
  The Hamilton Anxiety Rating Scale (HAMA) is a designed to assess symptoms of anxiety. Items are scored with a range of 0-4. A total score is then calculated of all items which can range from 0 to 54. A higher score is indicative of more anxiety symptoms, and a lower score post-tx is indicative of better outcome.
Beck Anxiety Inventory（BAI） | 1 months
  The Beck Anxiety Inventory (BAI) is a 21-item self-report questionaire that measures Anxiety symptoms. Each item is scored on a scale of 0-3, and items are summated to yield a total score. A higher score is indicative of greater symptoms of anxiety. Total scores may range between 0 and 63. A score greater than or equal of 8 is suggestive of clinically significant symptoms.
Mini-mental State Examination（MMSE） | 1 months
  The MMSE consists of 2 parts: language (time orientation (5 items), registration and attention) and performance (recall, response to written/verbal commands, sriting ability and reproduction of complex polygons); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement from baseline.
Montreal Cognitive Assessment Scale（MoCA） | 1 months
  The MoCA explores 8 cognitive domains: visuospatial/executive (score range form 0 to 5), naming(0-3), attention (0-5), language (0-3), abstraction(0-2), delayed recall(0-5), and orientation(0-6). The MoCA score was not corrected according to education level as advised by Gagnon and colleagues (2013). Its normal value was≥26 as proposed. A lower score indicates more severe cognitive impairment.
Named test of the Aphasia Battery of Chinese | 1 months
  The Aphasia Battery of Chinese(ABC) was compiled by Surong Gao et al in 1988 in accordance with the basic principles of aphasia inspection.It is mainly based on the Western Aphasia Battery (WAB), which has been developed through exploration and modification in combination with Chese national conditions and clinical experience.The named test is one of the subtest of the ABC.A total score is then calculated of all items which can range from 0 to 82. A higher score is indicative of worse outcome.
Similarity test | 1 months
  The similarity test includes 13 items scored with a range of 0-2. In each item, participants are given two words or concepts and have to describe how they are similar. A lower score indicates more severe abstract verbal reasoning and semantic knowledge impairment.
Symbol Digit modalities test（SDMT） | 1 months
  The Symbol Digit modalities test（SDMT) consists of nine digit-symbol pairs followed by a list of digits. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the 90 sec is measured.
Verbal fluency test（VFT） | 1 months
  The verbal fluency test is a kind of psychological test in which participants have to produce as many words as possible from a category in a given time (usually 60 seconds). A 60-second limit for responses within each category was allowed. Higher scores represent better performance.
Logical memory test（LMT） | 1 months
  The Logical Memory, subtest of the WMS-R is a standardized assessment of narrative episodic memory. A short story is orally presented, and the examinee is asked to recall the story immediately.
Delayed memory test（DMT） | 1 months
  Approximately 5 and 30 min later of the Logical memory test, recall of the story is again elicited, which is called delayed memory test.
Digit span test（DST） | 1 months
  In digit span test, participants must recall a series of numbers in order. A lower score indicates more severe working memory, attention, encoding and auditory processing impairment.
Ten point clock test | 1 months
  The ten point clock test is a reliable test of cognitive function. A total score is then calculated of all items which can range from 0 to 10. A higher score is indicative of better outcome.
Uniform Parkinson's Disease Rating Scale Ⅲ（UPDRSⅢ） | 1 months
  The motor section of the Unified Parkinson Disease Rating Scale (UPDRSⅢ) is covers the motor evaluation of disability and includes ratings for tremor, slowness (bradykinesia), stiffness (rigidity), and balance; part IV covers a number of treatment complications including ratings of involuntary movements (dyskinesias), painful cramps (dystonia), and irregular medication responses (motor fluctuations). It consists of 27 items, each are scored with a range of 0-4, with total score ranges from 0 to108. A higher score is indicative of more severe motor symptoms.
Modified Hoehn & Yahr scale（H-Y） | 1 months
  The Hoehn&Yahr scale is a commonly used system for describing how the symptoms of Parkinson's disease progress. It was originally published in 1967 in the journal Neurology by Melvin Yahr and Margaret Hoehn and included stages 1 through 5. Since then, a modified Hoehn&Yahr scale was proposed with the addition of stages 1.5 and 2.5 to help describe the intermediate course of the disease. A higher score is indicative of more severe movement impairment.
Activity of Daily Living Scale（ADL） | 1 months
  ADL was developed by Lawton and Brody in 1969.It consists of Physical self-maintenance Scale (PSMS) and Instrumental Activities of Daily Living Scale (IADL).It is mainly used to assess the daily life ability of the subjects. The total score below 14 points is indicative normal.More than 16 points is indicative functional decline.The highest score is 56.
Parkinson's Disease Questionnaire（PDQ-39） | 1 months
  The Parkinson's Disease Questionnaire is designed to address aspects of functioning and well-being for those affected by Parkinson's disease. Substantial evidence is available to suggest that the PDQ is reliable, valid, responsive, acceptable and feasible as the tool for the assessment of quality of life in Parkinson's disease patients. There are 39 questions in the long form Parkinson's Disease Questionnaire, with 8 discrete scales:mobility (10 items),activities of daily living (6 items),emotional well-being (6 items),stigma (4 items),social support (3 items),cognitions (4 items),communication (3 items),bodily discomfort (3 items) . Items are scored with a range of 0-4. A total score is then calculated of all items which can range from 0 to 156. A higher score is indicative of worse outcome.
Pittsburgh Sleep Quality Index (PSQI) | 1 months
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. A total score is then calculated of all items which can range from 0 to 21. A higher score is indicative of worse outcome.
Epworth Sleepiness Scale (ESS) | 1 months
  The Epworth sleepiness scale (ESS) is a self-administered questionnaire that's routinely used to assess daytime sleepiness. The person filling in the questionnaire rates how likely they are to doze off during the day in different situations. Each of the activities listed has an assigned score from 0 to 3 that indicates how likely a person is to fall asleep during the activity, and the total score can range from 0 to 24. A higher score is associated with increased sleepiness.
Parkinson's Disease Sleep Scale (PDSS-2) | 1 months
  The Parkinson's Disease Sleep Scale (PDSS-2) allows people with Parkinson's Disease to self-rate and quantify the level of sleep disruption being experienced. Each of the sleep disruption listed has an assigned score from 0 to 4 that indicates the sleep disruption frequency within a week, and the total score can range from 0 to 60. A higher score is associated with increased sleep disruption.

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Wang, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol